CLINICAL TRIAL: NCT04652336
Title: Randomized Controlled Trial Comparing the Effect of Ligamentum Teres Cardiopexy on de Novo GERD Post LSG
Brief Title: Study Comparing the Effect of Ligamentum Teres Cardiopexy on de Novo GERD Post LSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GEM Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GHC-16-OCT/2020
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: GERD
Keywords: de Novo GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSG (Active Comparator): This group will receive standard laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- LSG with LTC (Experimental): This group will receive LSG along with the novel LTC procedure
  Interventions: Procedure: ligamentum teres cardiopexy with sleeve gastrectomy

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — Comparator arm - will receive standard laparoscopic sleeve gastrectomy
  Arms: LSG
Procedure: ligamentum teres cardiopexy with sleeve gastrectomy — experimental arm - Ligamentum teres will be divided from umbilicus to up to umbilical fissure. The ligament will then be wrapped around lower esophagus and sutured.
  Arms: LSG with LTC

SUMMARY:
The aim of this study is to investigate the effect of ligamentum teres cardiopexy on incidence of de Novo GERD.

DETAILED DESCRIPTION:
Laparoscopic Sleeve Gastrectomy (LSG) is now the most commonly performed bariatric surgery world wide. The results of LSG on outcomes of GERD are conflicting. It has been reported to increase the severity of pre existing GERD and also to cause new onset GERD in considerable number of patients.

In this study the effect of adding a novel procedure i.e. ligamentum teres cardiopexy,(LTC) to regular LSG on occurence of de Novo GERD will be investigated. de Novo GERD has been found to occur in 20% of cases post LSG.

This study is a randomized, prospective, parallel group, controlled trial to compare the effect of LSG versus LSG with LTC on occurence of de Novo GERD.

This is a single center based trial, being conducted in GEM hospital and research center, Coimbatore, Tamil Nadu, India. The trial has been approved by GEM research ethics committee.

Investigators are planning to enroll patients who are not having any objective or subjective evidence of GERD. The participants will be optimized as per institutional bariatric surgery protocol. After complete evaluation and optimization, participants will be randomized by computer generated random numbers into either LSG or LSG with LTC group.

The demographic data, preoperative GERD - Q scores, 24 hour pH study, intra operative details will be recorded. Post operative details during each follow up will be recorded, which will include excess weight loss, GERD - Q scores. At 6 months follow up repeat 24 hour pH study will be done to assess the status of GERD objectively.

The trial duration is expected to be of 1 year where in investigators will be recruiting patients for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* candidate for bariatric surgery according to IFSO - APC guidelines
* No evidence (objective and subjective) of GERD

Exclusion Criteria:

* Presence of GERD either by history or by 24 hr pH study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-10 (Estimated); Primary Completion 2021-05-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
GERD | 6 months
  Subjective (Gastroesophageal Reflux Disease questionnaires - GERD - Q) and objective (24 hour pH study) measurement of occurence of GERD will be done GERD - Q - Score 0-2 denotes no GERD. Score more than or equal to 3 indicates presence of GERD 24 hr pH study - Demeester score more than 14.7 is indicative of presence of GERD

IPD SHARING:
Plan to Share IPD: Undecided